CLINICAL TRIAL: NCT02649673
Title: Phase Ib Dose-Escalation Study of LCL161 in Combination With Oral Topotecan for Patients With Relapsed/Refractory Small Cell Lung Cancer (SCLC) and Select Gynecologic Malignancies
Brief Title: LCL161 Plus Topotecan for Patients With Relapsed/Refractory Small Cell Lung Cancer and Select Gynecologic Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Clinical program was discontinued by Novartis
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI REFMAL 314
Record Dates: First submitted 2016-01-05; First posted 2016-01-07 (Estimated); Last update posted 2023-12-05 (Actual); Status verified 2022-06

CONDITIONS: Small Cell Lung Cancer; Ovarian Cancer
Keywords: lung carcinoma; topotecan; Hycamtin; ovarian neoplasms; LCL161; IAP inhibitors
MeSH Terms: conditions — Small Cell Lung Carcinoma; Ovarian Neoplasms; Lung Neoplasms | interventions — LCL161; Topotecan; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LCL161+topotecan+Pegylated GCSF (PEG-GCSF) (Experimental): Dose Escalation: Groups of 3-6 patients per dose level (DL) will initiate treatment in escalating doses until the maximum tolerated dose (MTD) is reached. MTD is defined as the highest combination of doses that results in dose-limiting toxicities for 2 of 6 patients per dosing group.
  * LCL161: orally, on Days 1, 8, 15 of each 21-day cycle. Maximum dose not to exceed 1200 mg/week.
  * topotecan: orally, for first 5 days of each 21-day cycle. Maximum dose not to exceed 2.3 mg/m2 per day.
  * Pegylated GCSF (PEG-GCSF) on-body injector (OBI) or daily GCSF (e.g. filgrastim) will be given according to institutional policy after Day 5 of topotecan. Because patients treated with topotecan are at high risk of developing febrile neutropenia, GCSF will be given in the prophylactic setting.
  Dose Expansion: 24 additional patients will be treated at the MTD in 2 cohorts (SCLC-12 patients; ovarian cancer-12 patients)
  Interventions: Drug: LCL161; Drug: Topotecan; Drug: Pegylated GCSF (PEG-GCSF)

INTERVENTIONS:
Drug: LCL161
Drug: Topotecan — Topotecan will also be administered orally. Patients in DL 1 will receive topotecan at 1.8 mg/m2 per day for the first 5 days of each 21-day cycle. Patients in DL 2 will receive topotecan at 2.3 mg/m2 per day for the first 5 days of each 21-day cycle. The maximum dose for topotecan will not exceed 2.3 mg/m2 per day in this study.
  Other Names: Hycamtin®
Drug: Pegylated GCSF (PEG-GCSF) — Pegylated GCSF (PEG-GCSF) (e.g. pegfilgrastim) on-body injector (OBI) or daily GCSF (e.g. filgrastim) will be given according to institutional policy after Day 5 of topotecan. Because patients treated with topotecan are at high risk of developing febrile neutropenia, GCSF will be given in the prophylactic setting.
  Other Names: pegfilgrastim

SUMMARY:
This trial will investigate the combination of two anti-cancer agents to treat patients with relapsed/refractory small cell lung cancer (SCLC) and ovarian cancers. Oral topotecan has US FDA approval for treating select gynecological cancers and SCLC. LCL161 is an investigational product that has been shown in clinical trials to work together with other anti-cancer agents. In this trial, investigators will determine the optimal dose of LCL161 and topotecan to administer to patients with relapsed/refractory SCLC and ovarian cancers, and examine the safety profile of the drug combination.

DETAILED DESCRIPTION:
This is an open-label, multicenter, non-randomized dose-escalation study of oral LCL161 administered in combination with oral topotecan. Topotecan is US FDA approved for treating metastatic ovarian cancer, stage IV-B cervical cancer, and small cell lung cancer (SCLC). LCL161, an investigational product, is an oral small-molecule antagonist of inhibitors of apoptosis proteins (IAPs). Preclinical data suggests that IAP antagonists work in synergy with other anti-cancer agents. This study is designed to evaluate the combination of these two agents in patients with SCLC and ovarian cancers where treatment with topotecan would be appropriate. The study will be conducted in 2 parts. In the dose-escalation part of the study, patients with relapsed/refractory SCLC and gynecologic malignancies will be eligible for enrollment to determine the optimal dose of the drug combination to be administered. Patients can continue treatment until disease progression or unacceptable toxicity. The dose-expansion part of the study is limited to patients with ovarian cancer and relapsed/refractory SCLC (2 cohorts with 12 patients each) to further assess safety and preliminary anti-tumor activity. Up to 52 patients are planned for enrollment at 3 centers in the U.S.

ELIGIBILITY:
Inclusion Criteria:

* Dose Escalation Portion: Must have histological diagnosis of relapsed/refractory SCLC or gynecological malignancy for which topotecan would be indicated.
* Dose Expansion Portion: Must have histological diagnosis of relapsed/refractory SCLC or ovarian cancer for which topotecan would be indicated.
* Patients must have evidence of recurrent epithelial ovarian, fallopian tube, or primary peritoneal cancer and must have previously received a platinum- / taxane-based chemotherapy regimen unless contraindicated. Only patients with platinum-resistant disease (recurrence < 6 months after platinum-based chemotherapy) are eligible.
* Patients with SCLC must have received platinum-based chemotherapy unless contraindicated.
* Patients must provide written informed consent prior to any screening procedures.
* Measurable or non-measurable (but evaluable) disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 (Eisenhauer et al. 2009)
* Required baseline laboratory status:
* Hemoglobin ≥90 g/L (9 g/dL)
* Platelets ≥100 x 109/L (100,000/mm3)
* Absolute neutrophil count (ANC) ≥1.5 x 109/L (1500/mm3)
* Serum total bilirubin ≤1.5 x the upper limit of normal (ULN) (in patients with known Gilbert Syndrome, a total bilirubin ≤3.0 x ULN, with direct bilirubin ≤1.5 x ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 x the ULN, except for patients with tumor involvement of the liver who must have ALT and AST ≤5 x ULN
* Creatinine clearance ≥ 50 mL/min, (measured by Cockcroft-Gault method):
* Aged ≥18 years
* Ability to swallow and retain oral medication
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.
* Life expectancy ≥12 weeks
* Male patients with female partners of childbearing potential and female patients of childbearing potential are required to use two forms of acceptable contraception, including one barrier method, during their participation in the study and for 6 months following last dose of study drug. Male patients must also refrain from donating sperm during their participation in the study.
* Ability to understand the nature of this study and comply with the study procedures and laboratory tests.

Exclusion Criteria:

* Patients with brain metastases may be enrolled if radiation and/or surgery have been completed and follow-up evaluation by computed tomography (CT) or magnetic resonance imaging (MRI) after 1 month demonstrates stable disease (SD), and the patient does not require corticosteroids or enzyme-inducing anti-epileptic medications for central nervous system disease. Patients with SCLC should have brain imaging performed within the last 2 months prior to study entry.
* More than 3 prior cytotoxic chemotherapy regimens given in the metastatic setting.
* Second-line ovarian cancer patients that are platinum-sensitive.
* Most recent chemotherapy ≤21 days and unresolved toxicities National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v4.03 Grade ≥2 (except alopecia)
* Use of an investigational drug ≤21 days or 5 half-lives (whichever is shorter) prior to the first dose of LCL161. For study drugs for which 5 half-lives is ≤21 days, a minimum of 14 days between termination of the study drug and administration of LCL161 is required
* Impairment of gastrointestinal function or gastrointestinal disease that may alter absorption of oral medications
* Major surgery ≤3 weeks or minor surgical procedures ≤7 days prior to study entry. No waiting is required following port-a-cath placement.
* Patients who are currently receiving chronic (>14 days) treatment with corticosteroids at a dose ≥10 mg of prednisone (or its glucocorticoid equivalent) per day, or any other chronic immunosuppressive treatment that cannot be discontinued prior to starting study drug
* Patients who are currently receiving treatment with agents that are metabolized solely through cytochrome P450 (CYP) 3A4/5 (CYP3A4/5) and have a narrow therapeutic index or are strong CYP2C8 inhibitors; or are receiving treatment with agents that carry a risk for QT prolongation and are CYP3A substrates. Caution should be used in patients taking other CYP2C8- or CYP3A4/5-interacting agents.
* New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities (see Appendix B), prolongation of the QTc interval to >450 msec for males or >470 msec for females on baseline electrocardiogram (ECG) per institutional standard or any of the following:
* History or presence of ventricular tachyarrhythmia
* Presence of unstable atrial fibrillation; patients with stable atrial fibrillation are eligible, provided they do not meet any of the other cardiac exclusion criteria.
* Clinically significant resting bradycardia (<50 bpm)
* Angina pectoris or acute myocardial infarction ≤3 months prior to starting study drug
* Other clinically significant heart disease (e.g., symptomatic congestive heart failure, uncontrolled arrhythmia or hypertension)
* Patients who are pregnant (positive beta-human chorionic gonadotropin [β-HCG]) or breastfeeding.
* Women of childbearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for at least 6 months after study treatment. Highly effective methods include:
* Total abstinence or
* Male partner or female sterilization or
* Combination of any two of the following (a+b or a+c or b+c):
* Use of oral, injected, or implanted hormonal methods of contraception
* Placement of an intrauterine device (IUD) or intrauterine system (IUS)
* Barrier methods of contraception: condom for male partner or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.

Note: Postmenopausal women are allowed to participate in this study. Women are considered post-menopausal and not of childbearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least 6 weeks ago. In the case of oophorectomy alone, a woman is considered to be not of childbearing potential only when her reproductive status has been confirmed by follow-up hormone level assessment.

* Wide field radiotherapy (including therapeutic radioisotopes such as strontium 89) administered ≤28 days or limited field radiation for palliation ≤7 days prior to starting study drug or has not recovered from side effects of such therapy
* Known diagnosis of human immunodeficiency virus, hepatitis B, or hepatitis C Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-03-23 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
The incidence of dose-limiting toxicities (DLTs) as a measure of safety and tolerability | 21 days (one cycle)
  The maximum tolerated dose (MTD) of the LCL161/topotecan combination is defined as the highest dose that results in dose-limiting toxicities (DLTs) for 2 of 6 patients during the first 21 days (1 cycle) of treatment, assessed using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.

SECONDARY OUTCOMES:
The incidence of acute and chronic treatment-emergent adverse events to further assess safety of the regimen | weekly for first 3 weeks then every 3 weeks thereafter, projected 6 months.
  The frequency and severity of AEs for all patients receiving at least one dose of treatment will be analyzed per NCI CTCAE v4.
Best overall response | every 6 weeks, projected 6 months
  Preliminary anti-tumor activity associated with combination treatment will be described using the best overall response recorded from start of treatment until disease progression, assessed per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Johnson, MD, Study Chair — SCRI Development Innovations, LLC
Locations (3):
- United States (3):
  - Florida Cancer Specialists-Sarasota, Sarasota, Florida
  - Oklahoma University Health Science Center/Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Tennessee Oncology PLLC, Nashville, Tennessee

REFERENCES:
- [Derived] Johnson ML, Patel MR, Aljumaily R, Jones SF, Burris Iii HA, Spigel DR. A Phase Ib Dose-Escalation Study of LCL161 Plus Oral Topotecan for Patients With Relapsed/Refractory Small Cell Lung Cancer and Select Gynecologic Malignancies. Oncologist. 2023 Jul 5;28(7):640-e559. doi: 10.1093/oncolo/oyad029. PMID 37129455